CLINICAL TRIAL: NCT05954208
Title: The Effect Of Visual Arts Group Therapy Based On Watson's Human Care Model On Perceived Social Support And Functional Recovery In Individuals With Schizophrenia
Brief Title: Vısual Arts Group Therapy Based On Watson's Human Care Model In Indıvıduals Wıth Schızophrenıa
Acronym: VAGT-WHCMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Nurcan Düzgün, Lecturer, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 78643
Record Dates: First submitted 2023-07-04; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia; Art Therapy; Social Support
Keywords: Schizophrenia; Visual arts therapy; Nursing model; Perceived social support; Functional recovery; Randomized controlled study
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VAGT-WHCM (Experimental): Vısual Arts Group Therapy Based On Watson's Human Care Model
  Interventions: Other: Vısual Arts Group Therapy Based On Watson's Human Care Model
- Control group (Active Comparator): Routine follow-up, treatment in the institution
  Interventions: Other: Ongoing treatment

INTERVENTIONS:
Other: Vısual Arts Group Therapy Based On Watson's Human Care Model — VAGT-WHCM was applied to the intervention group, consisting of six sessions, lasting 90 minutes on average, once a week in three groups.
  Arms: VAGT-WHCM
Other: Ongoing treatment — The control group participated only in the routine follow-up, treatment and practices in the institution.
  Arms: Control group

SUMMARY:
Purpose: This study was conducted to evaluate the effect of Visual Arts Group Therapy based on Watson's Human Care Model (VAGT-WHCM) on perceived social support and functional improvement in individuals with schizophrenia.

Design: This research was carried out as a randomized controlled experimental study with a pre-test-post-test and follow-up design, which is one of the quantitative research methods.

Method: The study was carried out in Yenimahalle Community Mental Health Center between December 2022 and January 2023. The sample of the study consisted of 67 individuals diagnosed with schizophrenia, including the intervention (n=34) and control group (n=33), who met the inclusion criteria and were determined by simple randomization method. VAGT-WHCM was applied to the intervention group, consisting of six sessions, lasting 90 minutes on average, once a week in three groups. The control group participated only in the routine follow-up, treatment and practices in the institution. The intervention and control groups were evaluated with the "Multidimensional Scale of Perceived Social Support (MSPSS)" and the "Functional Recovery Scale (FRS)" before therapy (pre-test), post-therapy (post-test), and one month later (follow-up). The CONSORT (Consolidated Standards of Reporting Trials) flowcart is used in this study.

Hypothesis:

H1-1: Visual arts group therapy has an effect on perceived social support by individuals with schizophrenia.

H1-2: Visual arts group therapy has an effect on the functional recovery levels of individuals with schizophrenia.

H1-3: The change in the perceived social support level of individuals with schizophrenia before and after visual arts group therapy is associated with the change in functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Meeting the diagnostic criteria for schizophrenia according to DSM-5 and being diagnosed with schizophrenia
* Being 18 years or older
* Being in remission (reported by the psychiatrist following the patient in the institution)
* Having medium and high level of insight (reported by the psychiatrist following the patient in the institution)
* Ability to read, understand and respond to instructions and data forms used

Exclusion Criteria:

* Having a diagnosis of a psychotic mental disorder in addition to the diagnosis of schizophrenia
* Using alcohol or psychoactive substances (reported by the doctor/nurse following the patient in the institution)
* Having a mental illness that makes cooperation impossible, such as mental retardation or dementia
* Having a serious physical illness such as cancer
* Being in an acute psychotic process
* Having visual, auditory, speech (verbal) and upper extremity defects
* Having participated in an art therapy program before
* Continuing any individual therapy or group therapy during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Perceived Social Support | Change from patients' perceived social support levels at two months
  The scale, which consists of a total of 12 questions, is evaluated in a 7-point Likert type. The participant chooses one of the options from 'Absolutely No' to 'Definitely Yes' in order to express the perceived support. It consists of three subscales, which are family, friend and personal support, which reflect the sources of support within the scale. The lowest total score that can be obtained from the scale is 12, and the highest score is 84. It is not the cut-off point of the scale, and the high score obtained from the scale indicates that the perceived social support is high.
Functional Recovery | Change from patients' functional recovery levels at two months
  The scale is a 5-point Likert-type scale consisting of 19 items. There are 5 evaluation levels for each item in the scale. Level 1 (absent) indicates the lowest level of improvement, while level 5 (excellent level) corresponds to the ideal level of functioning. It consists of Level 2 (partially present), Level 3 (have enough), Level 4 (almost fully present). High scores from the scale indicate high functionality, and low scores from the scale indicate low functionality. When you fall between the two levels, the lower level is selected. The maximum score that can be obtained from the scale is 95, and the minimum score is 19.The scale consists of 4 sub-dimensions. These are social functioning, health and treatment, daily living skills and occupational functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No